CLINICAL TRIAL: NCT01868412
Title: Comparison of Resin Salve and Medical Honey in Wound Care in Vascular Surgery Patients - A Prospective, Randomized and Controlled Clinical Trial
Brief Title: Resin Salve Versus Honey Treatment in Wound Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kuopio University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KUH15101075
Record Dates: First submitted 2013-05-08; First posted 2013-06-04 (Estimated); Last update posted 2016-01-18 (Estimated); Status verified 2016-01

CONDITIONS: Wound Healing; Wound Infection
Keywords: Wound healing; Wound infection; Resin salve; Medical honey
MeSH Terms: conditions — Wound Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Resin & honey (Experimental): Abilar 10% resin salve
  Interventions: Device: Abilar 10% resin salve
- Resin vs. honey (Active Comparator): Activon Tube 25 g
  Interventions: Device: Activon Tube 25 g

INTERVENTIONS:
Device: Abilar 10% resin salve — The resin salve may be spread directly onto the wound, after which the area is covered with a bandage suitable for local wound care. The bandage prohibits salve from moving away from the wound area. If the skin condition is more widespread or contains cavities or fistulae, the salve may be spread as a film with a thickness of at least 1 mm onto a gauze or gauze ribbon that is then used to fill the cavity or fistulae channel. Bandages are changed every 1-3 days, depending on the degree of infection and amount of wound secretion.
  Arms: Resin & honey
Device: Activon Tube 25 g — Wound care with the medical honey is carried out in the same manner than the resin salve treatment: honey may be spread directly onto the wound and the wound area is covered with a bandage suitable for local wound care. Similarly, if the skin condition is more widespread or wound contains cavities or fistulae, the medical honey may be spread as a film with a thickness of at least 1 mm onto a gauze or gauze ribbon that is then used to fill the cavity or fistulae channel. Bandages are changed every 1-3 days, depending on the severity of infection and amount of wound secretion.
  Arms: Resin vs. honey

SUMMARY:
In recent years, salve prepared from Norway spruce (Picea abies) resin and refined honey from manuka myrtle (Leptospermum scoparium), has successfully been used in medical context to treat both acute and chronic surgical wounds. The objective of this prospective, randomized and controlled clinical trial is to investigate healing rate and healing time of surgical wounds in patients, who have undergone peripheral vascular surgery, and whose complicated wounds are candidate for topical treatment with the resin or honey. In addition, factors contributing with delayed wound healing, antimicrobial properties, safety and cost-effectiveness of the resin salve and medical honey will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Infected of non-infected acute or chronic wound after vascular surgery.
* Need for topical wound care.
* Need for wound healing follow-up at the surgical outpatient department.

Exclusion Criteria:

* Life expectancy less than 6 months.
* Advanced malignant disease.
* Need for extensive surgical wound revision or skin transplantation.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-05; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Wound Healing | 6 months
  Healing rate of acute or chronic surgical wound within 6 months after vascular surgery (%).

SECONDARY OUTCOMES:
Contributors for Wound Healing | 6 months
  Contributors in terms of risk ratio (RR) to delayed wound healing.

OTHER OUTCOMES:
Other Pre-specified Outcome Measure | 6 months
  * Safety and compliance related with the resin salve or medical honey treatment.
  * Eradication rate of cultured pathogenic bacteria from wounds within 6 months.
  * Overall costs of resin salve and medical honey treatment within 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Tommi Auvinen, MD, Principal Investigator — Kuopio University Hospital
Locations (1):
- Kuopio University Hospital, Kuopio, Kuopio, Finland